CLINICAL TRIAL: NCT06914648
Title: The DRAGON PLC Trial - An International Multicenter Randomized Controlled Trial to Compare Combined Portal and Hepatic Vein Embolization (PVE/HVE) With PVE Alone in Primary Liver Cancers.
Brief Title: The Dragon PLC Trial (DRAGON-PLC)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL87590.0681.24
Record Dates: First submitted 2025-03-21; First posted 2025-04-06 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-02

CONDITIONS: Primary Liver Cancer; Hepatocellular Carcinoma (HCC); Cholangiocarcinoma
Keywords: Primary liver cancer; Future Liver Remnant; Liver regeneration; Portal Vein Embolization (PVE); Hepatic Vein Embolization (HVE)
MeSH Terms: conditions — Carcinoma, Hepatocellular; Cholangiocarcinoma

STUDY DESIGN:
Intervention Model Description: 1:1 Randomization between control and interventional group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Portal Vein Embolization (PVE) - control arm (Active Comparator): Portal Vein Embolization (PVE) alone
  Interventions: Procedure: Portal Vein Embolization
- Combined Portal and Hepatic Vein Embolization (PVE/HVE) - Interventional arm (Experimental): Combined Portal and Hepatic Vein Embolization (PVE/HVE)
  Interventions: Procedure: Portal Vein Embolization; Procedure: Hepatic Vein Embolization

INTERVENTIONS:
Procedure: Portal Vein Embolization — Description: Portal Vein embolization with Glue by a transhepatic approach
Procedure: Hepatic Vein Embolization — Hepatic Vein Embolization with Vascular plugs via a transjugular or transfemoral approach in the same session as the PVE procedure
  Arms: Combined Portal and Hepatic Vein Embolization (PVE/HVE) - Interventional arm

SUMMARY:
The goal of the DRAGON PLC clinical trial is to determine whether portal vein embolization (PVE) combined with hepatic vein embolization (HVE) improves resectability and overall survival in patients with initially unresectable primary liver cancer compared to standard PVE alone. This trial specifically focuses on patients with hepatocellular carcinoma and cholangiocarcinoma.

The main questions this trial aims to answer are whether combined PVE and HVE increases the proportion of patients who become resectable within 3 weeks and improves 5-year overall survival compared to PVE alone by enhancing liver hypertrophy.

Participants will:

* Undergo either standard PVE or combined PVE and HVE.
* Have regular imaging to assess liver resectability.
* Be monitored for survival outcomes up to 5 years after intervention.

DETAILED DESCRIPTION:
Primary liver cancer (PLC) is the third most common cause of cancer death worldwide. Surgical resection is the mainstay for a curative approach as contemporary chemotherapy and immune-based therapies only lead to a median survival of 10-14 months. A complete surgical resection increases the median survival to 42 months (range 32-52 months). However, PLC is mainly diagnosed at an advanced stage and >70% of PLC patients are ineligible for an immediate surgical approach. There are different reasons that make a patient ineligible for surgery, one important reason is the risk of liver failure after the surgery due to a small remnant liver.

This study aims to improve the oncological, radiological and surgical strategy to allow more patients to undergo liver resection safely, to improve quality of life and to extend overall survival at acceptable costs.

Adequate function of the future liver remnant (FLR) is a prerequisite for surgical resectability. This is necessary in order to avoid liver failure after surgery, a major cause of morbidity (38%) and mortality (27%). To mitigate this risk, regenerative strategies based on preoperative calculation of the FLR volume and function are essential. Patients with technically resectable disease but predicted insufficient FLR volume or function are referred to as primarily unresectable or potentially resectable (PU/PR). These patients can undergo strategies that capitalize on the regenerative capacity of the liver which aim to preoperatively increase the FLR volume and function in order to allow surgery. Many of the patients that are primarily unresectable due to an insufficient FLR can become ultimately and safely resectable after the induction of adequate FLR-hypertrophy by the current standard, portal vein embolisation (PVE). However, 25% of patients do not show sufficient FLR growth after PVE and are unable to safely undergo resection. A new approach has been developed to improve this. Combined portal and hepatic vein embolisation (PVE/HVE) has great promise in terms of increasing FLR growth, resection rate (RR), safety and potentially, overall survival. Establishing PVE/HVE as the new standard could result in increased survival and a better quality of life (QoL) for patients.

ELIGIBILITY:
Inclusion Criteria:

* PLC diagnosis, specifically iCCC, pCCC, and HCC;
* Requiring PVE due to an FLR volume is <30% in normally functioning livers, <40% in livers with potentially impaired function e.g. resulting from prior systemic therapy induction or bile duct colonization / transpapillary biliary drainage, or <50% in livers with severely impaired function resulting from liver cirrhosis (max. Child Pugh A5) OR function on hepatobiliary scintigraphy (HEBIS) is < 2.7 %/min/m2;
* Age ≥ 18 years;
* Able to understand the trial and provide informed consent.

Exclusion Criteria:

* Liver cirrhosis with a Child-Pugh score of B or C;
* Presence of portal hypertension;
* Presence of cholangitis;
* Pregnant women;
* Premenopausal females not able/willing to commit to contraception (specifically long-acting reversible contraception or hormonal contraception);
* Patients unresectable due to prohibitive comorbidities (decision made by local multidisciplinary team);
* Patients with hepatic malignancies other than iCCC, pCCC or HCC;
* PVE/HVE anatomically not feasible;
* Any patient with non-resectable or non-ablatable extrahepatic metastatic disease.
* Unable to understand the study information, study instructions and give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 358 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2032-11-15 (Estimated); Study Completion 2032-11-15 (Estimated)

PRIMARY OUTCOMES:
Resectability 3 weeks after embolisation | 3 weeks
  The FLR is considered sufficient for resection 3 weeks after embolisation. Definition resectable: Patients are deemed resectable if the FLR is ≥30% in normally functioning livers, ≥40% in livers with potentially impaired function (e.g. resulting from prior systemic therapy or bile duct colonization / transpapillary biliary drainage), or ≥50% in livers with severely impaired function resulting from liver cirrhosis (max. Child Pugh A5) OR for any FLR volume, function on hepatobiliary scintigraphy is > 2.7 %/min/m2
Overall survival | 5 years
  survival data will be recorded up to 5-years

CONTACTS AND LOCATIONS:
Locations (55):
- United States (5):
  - Yale School of Medicine Hospital, New Haven, Connecticut
  - Rush University Medical Center, Chicago, Illinois
  - Mayo Clinic, Rochester, Minnesota
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
- Monash Medical Center, Melbourne, Australia
- Austria (2):
  - Medical University of Vienna, Vienna, Vienna
  - Social Center South, Vienna, Vienna
- Belgium (9):
  - Erasmus Hospital, Brussels, Brussels Capital
  - UZ Antwerpen, Antwerp, Edegem
  - UZ Gent, Ghent, Gent
  - CHU Liège, Liège, Liège
  - CHU-UCL Namur site Godinne (UCLouvain), Yvoir, Namen
  - Cliniques Universitaires Saint Luc, UCLouvain, Brussels
  - Jessa Hospital, Hasselt
  - UZ Brussel, Jette
  - AZ Groeninge Hospital Kortrijk, Kortrijk
- Canada (14):
  - Foothills Medical Center, Calgary, Alberta
  - Vancouver General Hospital, Vancouver, British Columbia
  - Queen Elizabeth II Health Sciences Center, Halifax, Nova Scotia
  - Juravinski Hospital and Cancer Centre, Hamilton, Ontario
  - Kingston Health Sciences Centre, Kingston, Ontario
  - London Health Sciences Centre, London, Ontario
  - St. Joseph's Health Centre, Toronto, Ontario
  - Sunnybrook Hospital, Toronto, Ontario
  - University Health Network/TGH, Toronto, Ontario
  - Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec
  - Centre Hospitalier de l'Université de Montréal, Montreal
  - McGill University Health Centre, Montreal, Montreal
  - L'Hopital d'Ottawa, Ottawa
  - Royal University Hospital, Saskatoon
- Germany (3):
  - Universitätklinikum Köln, Cologne
  - Universitätklinikum Dresden, Dresden
  - Universitätklinikum Hannover, Hanover
- Ospedale San Raffaele, Milan, Italy
- Netherlands (5):
  - Maastricht Universitair Medisch Centrum+, Maastricht, Limburg
  - Amsterdam UMC, location VUMC, Amsterdam, North Holland
  - Maxima Medisch Centrum, Eindhoven
  - Universitair Medisch Centrum Groningen, Groningen
  - Leiden Universitair Medisch Centrum, Leiden
- University Hospital Oslo, Oslo, Norway
- Sweden (2):
  - University Hospital Linköping, Linköping
  - Karolinska University Hospital Stockholm, Stockholm
- Switzerland (6):
  - Cantonal Hospital Winterthur, Winterthur, Canton of Zurich
  - Claraspital Basel, Basel
  - Universitätsspital Basel, Basel
  - CHUV - Lausanne University Hospital, Lausanne
  - Hirslanden Klinik St. Anna, Lucerne
  - Hirslanden Klinik, Zurich
- United Kingdom (6):
  - Belfast Health and Social Care Trust, Belfast
  - Queen Elizabeth Hospital, Birmingham
  - Aintree University Hospital, Liverpool
  - Kings college Hospital, London
  - Oxford University Hospitals NHS Foundation Trust, Oxford
  - University Hospital Southampton, Southampton

IPD SHARING:
Plan to Share IPD: Yes
Upon reasonable request
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After publication
Access Criteria: Proposal accepted by the DRAGON Collaborative Scientific Committee

REFERENCES:
- See also: Related Info — https://www.dragontrial.com/